CLINICAL TRIAL: NCT03271645
Title: Internet-delivered Interventions for Stress, Anxiety and Depression in the Workplace
Acronym: iCBT@Work
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: logistics
Sponsor: Silver Cloud Health (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: iCBT@Work
Record Dates: First submitted 2017-08-24; First posted 2017-09-05 (Actual); Last update posted 2018-09-11 (Actual); Status verified 2018-09

CONDITIONS: Depression; Anxiety; Stress
Keywords: Depression; Anxiety; Stress; Internet-delivered interventions
MeSH Terms: conditions — Depression; Anxiety Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Space from depression (Experimental): Space from depression is an 8 module CBT-based intervention.
  Interventions: Behavioral: Space from Depression
- Space from Anxiety (Experimental): Space from anxiety CBT is an 8 module CBT-based intervention.
  Interventions: Behavioral: Space from Anxiety
- Space from stress (Experimental): Space from stress CBT is an 8 module CBT-based intervention.
  Interventions: Behavioral: Space from Stress
- Face-to-face counselling (Active Comparator): Face-to-face counselling
  Interventions: Behavioral: Face-to-face counselling

INTERVENTIONS:
Behavioral: Space from Depression — The structure and content of the programme modules follow evidence-based principles of CBT for the treatment of depression and anxiety (NICE, 2006, 2011, 2014). The treatment comprises cognitive, emotional and behavioural components. The treatment is delivered on a Web 2.0 platform using media-rich interactive content. Each module is structured in an identical way and incorporates introductory quizzes, videos, informational content, interactive activities, as well as homework suggestions and summaries. In addition, personal stories and accounts from other clients are incorporated into the presentation of the material.
  Arms: Space from depression
Behavioral: Space from Anxiety — The structure and content of the programme modules follow evidence-based principles of CBT for the treatment of depression and anxiety (NICE, 2006, 2011, 2014). The treatment comprises cognitive, emotional and behavioural components. The treatment is delivered on a Web 2.0 platform using media-rich interactive content. Each module is structured in an identical way and incorporates introductory quizzes, videos, informational content, interactive activities, as well as homework suggestions and summaries. In addition, personal stories and accounts from other clients are incorporated into the presentation of the material.
  Arms: Space from Anxiety
Behavioral: Space from Stress — The structure and content of the programme modules follow evidence-based principles of CBT for the treatment of depression and anxiety (NICE, 2006, 2011, 2014).The treatment is delivered on a Web 2.0 platform using media-rich interactive content. Each module is structured in an identical way and incorporates introductory quizzes, videos, informational content, interactive activities, as well as homework suggestions and summaries. In addition, personal stories and accounts from other clients are incorporated into the presentation of the material.
  Arms: Space from stress
Behavioral: Face-to-face counselling — Face-to-face counselling
  Arms: Face-to-face counselling

SUMMARY:
The research will utilise an open feasibility parallel groups trial to examine the impact of novel internet-delivered cognitive behavioural therapy (CBT) interventions for stress, anxiety, and depression compared to treatment as usual (face to face counselling and psychotherapy) in an employment context. Participants will consist of employees accessing services provided by employee assistance programmes (EAP) provided at the European headquarters of a large technology organisation.

DETAILED DESCRIPTION:
Participants will be recruited for the online intervention through either self-referral or a referral from one of the counsellors or GPs at the onsite well-being service centre. Participants in the face-to-face group will be recruited by referral from a member of the EAP; those on the waiting list for face-to-face services provided by the EAP will be approached to participate in the research. At baseline, participants in both the online and the face-to-face groups will complete sociodemographic information, the PHQ-4, PSS-4, the HPQ-SF, as well as an assessment of risk using question 9 from the PHQ-9. Eligible participants in the online intervention group will be offered one of three internet-delivered CBT interventions (Space from Stress, Space from Anxiety, Space from Depression). Participants attending the onsite EAP counselling service will receive 8 sessions of counselling.

Risk Assessment

Participants will be screened at baseline for risk. This assessment will be conducted through the response to question 9 on the PHQ-9, in which respondents are requested to indicate how often they have been bothered by "thoughts that you would be better off dead or of harming yourself in some way" rated on a 4-point Likert scale, with 0 indicated "not at all", 1 = "several days", 2 = "more than half the days", 3 = "nearly every day". Any participant who scores > 1 will be automatically prompted to answer additional questions to qualify the level of risk indicated. These questions include "Do you have any current plans to end your life?", "Have you made any actual preparations towards ending your life?" answered in a simple "yes/no" format and "how likely is it that you will act on these thoughts or plans to end your life" rated on a 0=10 scale with 0 indicating "I would never do this" and 10 indicating "I am definitely going to do this". Participants are also asked an open-ended question about their protective factors "what is stopping you from acting on these thoughts?". If any risk to self or others is highlighted, the participant will be immediately provided with crisis contact numbers (GP Out of Hours, Samaritans, Aware, Pieta House, Women's Aid, Amen) through the platform, and encouraged to contact these services directly if they feel in crisis. In addition, participants who indicate risk at baseline will be recommended that they contact the onsite GP or one of the counsellors at the onsite wellness centre. Those who exceed the cut-off score for risk ( >1 PHQ-9 Question 9) on the screening questions will not be eligible to participate in the study and will be able to access support from the onsite GP and /or the counselling team at the onsite wellness centre.

During the course of the trial, all supporters who are trained mental health practitioners will remain alert for indications of risk and will escalate concerns within the established supervision governance structure in an appropriate time frame.

During treatment, participants in both the online interventions and the face-to-face intervention will complete the PHQ-4 and PSS-4. At the end of the treatment, participants will be asked to complete the PHQ-4, PSS-4, SAT, and the HPQ-SF. These measures will also be completed at 4-months follow-up. A mixed-method approach will be used to include quantitative and qualitative analysis of symptom severity, work performance, and user satisfaction.

Each of the online interventions (Space from Depression, Space from Anxiety, Space from Stress) consists of 8 modules of internet-delivered CBT, delivered over an 8-week period. Participants will be assigned a supporter who will provide weekly post-session feedback on progress and exercises.

Support for this trial will be provided by Nuffield Health clinical support services. Nuffield Clinical Support Services is an established clinical service that provides support through Nuffield Health's Employee Assistance Programmes. The service is composed of British Association of Behavioural and Cognitive Psychotherapists (BABCP) accredited cognitive behavioural psychotherapists. They also have a small group of psychological well-being practitioners who are also British Association of Behavioural and Cognitive Psychotherapists (BABCP) accredited or currently in supervised training for accreditation. Each supporter will provide post-session feedback of between 10 and 15 minutes per participant per session.

Schedule of Assessment:

Participants will complete the primary and secondary outcome measures at baseline. Thereafter, they will complete the PHQ-4 and PSS-4 at each counselling or online review session. Once participants have completed treatment, they will be contacted to complete both the primary and secondary outcome measures. Satisfaction with treatment will be measured post-treatment at 4-month follow-up, where participants will complete the PHQ-4, PSS-4 and HPQ-SF.

Data analysis:

The feasibility of Internet-delivered interventions for stress, anxiety and depression as part of the organization's EAP will be evaluated based on participant recruitment, enrollment and retention rates.

Effectiveness over time of Internet-delivered interventions for the treatment of stress, anxiety and depression will be determined independently using linear mixed models. Stress severity will be measured using PSS-4 scores, depression and anxiety severity using PHQ-4 scores. In addition, sociodemographic characteristics will be assessed at baseline and factors significantly associated with treatment groups incorporated in the analysis model if required.

The impact of an internet-delivered intervention on workplace absence and job performance will be determined through the collection of HPQ-SF measures pre-treatment, immediately post-treatment and at 4-month follow-up. HPQ-SF absenteeism and presenteeism scores will be analysed using repeated measures ANOVA to detect differences at each time point.

Employee satisfaction with an internet-delivered intervention will be assessed in the Satisfaction with Treatment Questionnaire. Quantitative and qualitative measures of satisfaction will be summarised using descriptive statistics.

Internet-delivered intervention group:

Registered employees of the company will be eligible to participate in this study and will be recruited through the services their EAP provide. Participants may also be referred to the internet-delivered intervention by their general practitioner or other mental health professionals within the EAP. Interested participants will be able to log on to the SilverCloud Platform, where they can read the participant information sheet. Participants in the face-to-face group will be given a hard copy of the participant information sheet. This will detail what is involved with the study, the procedure, and how to proceed. Should participants agree to take part in the research, they will be requested to indicate their informed consent digitally. Participants will then complete the baseline measures. Participants excluded at this stage based on their risk assessment scores will be directed to the appropriate services within the EAP, for example, to the GP or face-to-face counselling services.

Using computer algorithms to score screening instruments at baseline, participants will be automatically provided with feedback on their measures (e.g. your scores indicate you may be experiencing moderate symptoms of depression). This feedback consists of informing the participant of their overall score for each measure and highlight the individual as the expert in their own life. All participants in the Internet-delivered intervention group will make an informed decision on choosing one of the three programmes, based on the combination of scores from the depression, anxiety, and stress scales. Participants will then self-select one of the three programmes: Space from Depression, Space from Anxiety, Space from Stress.

Each participant in the Internet-delivered intervention group will be assigned a supporter who will monitor participant's progress throughout the trial. Once a participant begins their chosen programme, they will receive a message from their supporter at their first log-in. This message welcomes them to the programme, highlights aspects of it and encourages them in the use of it. Weekly, supporters will log in and review participants progress, leaving feedback for them and responding to the work they have completed. Supporters will be BABCP accredited cognitive behavioural psychotherapists and psychological well-being practitioners who are also BABCP accredited or currently in supervised training for accreditation, provided by Nuffield Health EAP clinical support services. Each supporter will provide post-session feedback of between 10 and 15 minutes per participant per session.

Face to face counselling/psychotherapy group:

Once the trial starts, those beginning face-to-face services will be approached to participate in the research by a member of the EAP. Those who wish to participate will then sign a paper/ digital on iPad consent form and will complete measures at baseline and post-treatment, as per the schedule of assessment. Risk will be monitored by the clinician responsible for the participant.

The study is an open feasibility trial that uses standard instruments to assess symptoms of anxiety, depression and stress and adjustment psychopathology. It does this using reliable and valid instruments, including:

Patient Health Questionnaire (PHQ-4) a self-report measure of depression and anxiety that has been widely used in screening, primary care, and research. The PHQ-4 items reflect the diagnostic criteria for depression outlined by the Diagnostic and Statistical Manual of Mental Disorders, Fourth Edition - Text Revision (DSM-IV-TR).

Perceived Stress Scale (PSS-4): a self-report measure of non-specific perceived stress. Based on Lazarus's transactional model of stress respondents rate how unpredictable, uncontrollable, and overloaded they appraise their life to be. Items are answered on a 5-point Likert scale (0= never, 1=almost never, 2=sometimes, 3=fairly often, 4=very often) referring to the past month.

Health and Work Performance Questionnaire - Short Form: a brief self-report measure designed to estimate the workplace costs of health difficulties in two domains: absenteeism and reduced job performance. Validation studies have demonstrated significant correlations between self-reported HPQ scores and archival pay roll and performance assessments. The HPQ has been demonstrated to be valid, reliable and sensitive to change and recommended for use in Internet-delivered environments.

Satisfaction with Treatment (SAT) Questionnaire: includes nine quantitative items rated on a scale from 0 to 4 (e.g., How did this online treatment compare to previous treatments? 0 = 'Much better' to 4 = 'Not at all good'). The Satisfaction with Treatment questionnaire also contains two qualitative questions asking participants to describe what they liked most and least about the Internet-delivered intervention.

ELIGIBILITY:
Inclusion Criteria:

* All participants will be 18+ years of age.

Exclusion Criteria:

* Suicidal intent/ideation: score >1 on PHQ-9 question 9.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2018-09-11 (Estimated); Primary Completion 2019-03-01 (Estimated); Study Completion 2019-06-01 (Estimated)

PRIMARY OUTCOMES:
PHQ-4 | Up to 4-months
  Patient health Questionnaire
PSS-4 | Up to 4-months
  Perceived Stress Scale-4 (PSS-4)

SECONDARY OUTCOMES:
Health and Work Performance Questionnaire (HPQ-SF) | Up to 4-months
  Health and Work Performance Questionnaire
Satisfaction with Treatment Questionnaire (SAT) | 8 weeks
  Satisfaction with Treatment Questionnaire (SAT)

CONTACTS AND LOCATIONS:
Overall Officials: Derek Richards, PhD, Principal Investigator — SilverCloud Health
Locations (1):
- Multinational Technology Industry European HQ, Cork, Ireland

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Kroenke K, Spitzer RL, Williams JB. The PHQ-9: validity of a brief depression severity measure. J Gen Intern Med. 2001 Sep;16(9):606-13. doi: 10.1046/j.1525-1497.2001.016009606.x. PMID 11556941
- [Background] American Psychiatric Association. Diagnostic and statistical manual of mental disorders (DSM-IV-TR). 4th ed. Washington D.C.: American Psychiatric Association.; 2000.
- [Background] Cohen S, Williamson G. Perceived stress in a probability sample of the United States. In: S. Spacapan, Oskamp S, editors. The social psychology of health. Newbury Park, CA: Sage; 1988.
- [Background] Cohen S, Kamarck T, Mermelstein R. A global measure of perceived stress. J Health Soc Behav. 1983 Dec;24(4):385-96. No abstract available. PMID 6668417
- [Background] Kessler R, Petukhova M, McInnes K. World Health Organization Health and Work Performance Questionnaire (HPQ). HPQ Short Form (Absenteeism and Presenteeism Questions and Scoring Rules) Harvard Medical School. 2007.
- [Background] Kessler RC, Barber C, Beck A, Berglund P, Cleary PD, McKenas D, Pronk N, Simon G, Stang P, Ustun TB, Wang P. The World Health Organization Health and Work Performance Questionnaire (HPQ). J Occup Environ Med. 2003 Feb;45(2):156-74. doi: 10.1097/01.jom.0000052967.43131.51. PMID 12625231
- [Background] Kessler RC, Ames M, Hymel PA, Loeppke R, McKenas DK, Richling DE, Stang PE, Ustun TB. Using the World Health Organization Health and Work Performance Questionnaire (HPQ) to evaluate the indirect workplace costs of illness. J Occup Environ Med. 2004 Jun;46(6 Suppl):S23-37. doi: 10.1097/01.jom.0000126683.75201.c5. PMID 15194893
- [Background] Richards D, Timulak L. Satisfaction with therapist-delivered vs. self-administered online cognitive-behavioural treatments for depression symptoms in college students. British Journal of Guidance & Counselling. 2012;41(2):193-207
- See also: SilverCloud website — http://www.silvercloudhealth.com